CLINICAL TRIAL: NCT03987971
Title: Acupuncture on GB26 to Treat Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wenzhou Medical University (Other)
Collaborators: Qingtian People's hospital (Unknown)
Responsible Party: Principal Investigator, Tang Lewei, Principal Investigator, Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GB264LBP
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Chronic Low-back Pain
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Deep acupuncture on GB26 (Experimental)
  Interventions: Other: acupuncture
- Superficial acupuncture on GB26 (Sham Comparator)
  Interventions: Other: acupuncture
- waiting list (No Intervention)

INTERVENTIONS:
Other: acupuncture — Acupuncture on GB26, every other day, 3 times a week, 2 weeks in total.
  Arms: Deep acupuncture on GB26; Superficial acupuncture on GB26

SUMMARY:
This study evaluates the effecacy of acupoint GB26 based acupuncture treatment in patients with chronic low back pain. Half of the participants will partake in a 2-week acupuncture intervention, while the other half will receive a placebo treatment. The investigators hypothesize that acupuncture on GB26 reduces disability and pain more than the control intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults (both male and female) with non-specific low back pain for more than three months.
* Age range: between 20 and 60 years.
* Willingness of the patient to participate in the study, and written informed consent signed and personally dated by the patient.
* Chronic non-specific low back pain clinically diagnosed as repeated lumbar sourness and swelling pain or a chronic progressive process, accompanied by (i) X-ray examination to exclude lumbar vertebrate fractures, spondylolysis, spondylolisthesis and severe osteoporosis, and/or (ii) MRI with normal signal or low nucleus pulposus signal.

Exclusion Criteria:

* Age less than 20 or greater than 60 years
* Specific causes of back pain (e.g., cancer, fractures, spinal stenosis, infections)
* Complicated back problems (e.g., prior back surgery, medico-legal issues)
* Possible contraindications for acupuncture (e.g., coagulation disorders, cardiac pacemakers, pregnancy, seizure disorder), and conditions that might confound treatment effects or interpretation of results (e.g., severe fibromyalgia, rheumatoid arthritis)
* Conditions making treatment difficult (e.g., paralysis, psychoses, or other severe psychiatric problems based on the judgment of a physician investigator and/or a T score >60 on the psychological assessments performed during Session 1)
* Prior acupuncture treatment for back pain; 1 year minimum for any other condition.
* The intent to undergo surgery during the time of involvement in the study.
* History of cardiac, respiratory, or nervous system disease that, in the judgment of a physician investigator, precludes participation in the study because of a heightened potential for adverse outcome (e.g., asthma, claustrophobia)
* Presence of any contraindications to MRI scanning (e.g., cardiac pacemaker, metal implants, fear of closed spaces, pregnancy)
* Active substance abuse disorders within the last 24 months, based on subject self-report
* Radicular knee pain extending below the knee

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Change in Numerical Rating Scale (NRS) score | Change from baseline NRS score at 1 weeks, 2 weeks, 4 weeks and 12 weeks
  The NRS will ask patients to rate their pain intensity on an 11-point scale where 0 indicates no pain and 10 indicates worst imaginable pain
Change in Oswestry Low Back Pain Disability Questionnaire (OLDPDQ) score | Change from baseline NRS score at 1 weeks, 2 weeks, 4 weeks and 12 weeks
  The OLDPDQ score is considered the 'gold standard' of low back functional outcome tools. The questionnaire is composed of ten sections (addressing pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life and travelling); for each section the possible score is 5 and, thus, the total possible score is 50. The final score is calculated as [(sum of individual scores) / 50] *100 (%), and is interpreted as minimal disability (0% to 20%), moderate disability (21% to 40%), severe disability (41% to 60%), crippled (61% to 80%) or patients are either bed-bound or exaggerating their symptoms (81% to 100%).